CLINICAL TRIAL: NCT05558748
Title: "Comparison of Analgesic Effects of USG-Guided Caudal Versus Ilioinguinal/Iliohypogastric Nerve Block Techniques for Inguinal Surgeries in Children, a Randomized Controlled Trial."
Brief Title: "Comparison of USG-Guided Caudal Versus Ilioinguinal/Iliohypogastric Nerve Block for Pediatric Inguinal Surgeries"
Acronym: CAUCIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MREC#2919
Record Dates: First submitted 2022-09-25; First posted 2022-09-28 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-09

CONDITIONS: Analgesia; Inguinal Surgery; Undescended Testes; Hydrocele; Torsion Testis; Varicocele; Ilioinguinal Nerve Block
Keywords: inguinal surgery; caudal anesthesia; nerve block; inguinal hernia; postoperative pain
MeSH Terms: conditions — Agnosia; Cryptorchidism; Testicular Hydrocele; Spermatic Cord Torsion; Varicocele; Hernia, Inguinal; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The patients will be randomized using a computer-generated sequence to one of the two intervention groups: USG-guided Caudal block and USG-guided Ilioinguinal/Iliohypogastric block. There will be no crossover.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant (patient) and the outcome assessor will be masked. Whereas the investigator who performs the block will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric patients undergoing inguinal surgeries with USG-guided Caudal block. (Active Comparator): All pediatric patients (6 months to 12 year) posted for inguinal surgery under general anesthesia with USG-guided Caudal block for analgesia
  Interventions: Procedure: USG-guided Caudal block
- Pediatric patients undergoing inguinal surgeries with USG-guided Ilioinguinal/Iliohypogastric block. (Active Comparator): All pediatric patients (6 months to 12 year) posted for inguinal surgery under general anesthesia with USG-guided Ilioinguinal/Iliohypogastric block for analgesia
  Interventions: Procedure: USG-guided Ilioinguinal/Iliohypogastric block

INTERVENTIONS:
Procedure: USG-guided Caudal block — USG-guided Caudal block after general anesthesia
  Arms: Pediatric patients undergoing inguinal surgeries with USG-guided Caudal block.
Procedure: USG-guided Ilioinguinal/Iliohypogastric block — USG-guided Ilioinguinal/Iliohypogastric block after general anesthesia
  Arms: Pediatric patients undergoing inguinal surgeries with USG-guided Ilioinguinal/Iliohypogastric block.

SUMMARY:
This study is designed to compare the analgesic effectiveness of caudal analgesia to ilioinguinal regional analgesia techniques in children undergoing inguinal surgeries. Both techniques will be done under ultrasound gaudiness, using the same local anesthesia. 128 patients will be included in this study, 64 for each technique. This study aims to know the best regional analgesia technique in children undergoing inguinal surgeries, reduction in rescue analgesia postoperatively, postoperative length of stay, and early resumption of postoperative activity.

The patients will be followed up 30 minutes after the end of anesthesia in PACU, postoperatively in Ward at 2 Hours, 3 hours, 6 hours from the end of anesthesia, and or at the time of discharge from the ward & on days 2 and 7. Patient privacy and safety will be respected at all times. An interim analysis will be done after recruiting 25% of cases (16 cases) in both arms. Once the sample size is reached, the data will be sent for statistical analysis with coded patient identity.

Based on study findings, the practice will be optimized with the aim of improvement in pain relief, reduction in opioid requirements, and enhanced recovery after surgery (ERAS), reducing the bed occupancy time in the hospital.

DETAILED DESCRIPTION:
Introduction Inguinal surgeries are commonly performed in children. Pain is a dreaded side effect of any surgery and should be adequately assessed and treated. It has been shown that even minor procedures can cause significant pain in children.

1. Assessment of adequate analgesia is complex in children. Inadequate analgesia can cause neurological, metabolic, pulmonary, and other bodily effects.
2. Postoperative analgesia for inguinal surgeries can be provided with caudal and ilioinguinal/iliohypogastric nerve blocks. These techniques are safe and reduce the requirement for opioids postoperatively. This can help in early discharge from the hospital and faster resumption of daily activities.

   The caudal block involves an injection of local anesthetic agents into the caudal space. The caudal space is the sacral portion of epidural space involving needle penetration of sacrococcygeal ligament covering sacral hiatus. This block is commonly done to provide analgesia for urogenital, rectal, and inguinal surgeries. This block was primarily performed as a blind technique. The onset of action is typically in 8.8 minutes, as per NYSORA guidelines. Fortunately, serious complications occur infrequently. Potential complications include epidural abscess, meningitis, epidural hematoma, dural puncture, post-dural puncture headache, subdural injection, pneumocephalus, air embolism, back pain, and intracranial hypotension headache after uncomplicated caudal epidural injection. Ilioinguinal/iliohypogastric nerve block is commonly performed for inguinal surgeries. This nerve penetrates the transversus abdominis muscle above the iliac crest and supplies the muscle, and provides cutaneous innervation to the skin of the scrotum and adjacent thigh. This block is known to abolish pain following inguinal surgeries in the pediatric population effectively.

   The primary objective of the study is to find a better analgesia technique out of caudal and ilioinguinal/iliohypogastric blocks. The secondary objective is to compare the reduction in the use of rescue analgesics and find a technique that provides earlier resumption of activities.

   Methods:

   Study type: Randomized Controlled Trial, with 2 parallel arms. Blinding: Double blinding: The patient, as well as the postoperative assessor, will be blinded.

   Crossover: Nil Study duration: Prospective for 6-12months depending on the case recruitment rate.

   Number of groups: 2 Sample size: 128 patients (64 patients for each technique ) Target follow-up duration: Intraoperative period, at 30 minutes after arrival and before discharge from PACU, postoperatively in Ward at 2 Hours, 3 hours, 6 hours, and or at time of discharge from the ward and at home on day 2 and day 7.

   Study population Sample size The estimated sample size is 128 (64 in each group). The estimation was based on the anticipated effect size (medium, Cohen's d= 0.5) for the difference in the post-operative pain score between caudal and ilioinguinal block methods. The power was set at 80%, and the alpha error was set at 5%. The allocation ratio will be 1:1. The software used for the sample size calculation is G*Power version 3.1.9.7

   Method:

   An appropriate population posted for surgery will be approached as per eligibility criteria, will be approached. An explanation of the study will be done in comprehensive language. The patient's rights will be explained to the patient/relatives. Informed consent will be taken on the consent form. The patient will then be randomized into 3 age-stratified groups (6 months up to 3 years, 3 years onwards to 6 years, and 6 years onwards to 12 years). Each patient will be randomized to group A or B according to the computer-generated stratified age group block randomization sequence. The randomization sequence will be kept locked with a password-protected file. It will be accessed at the time of randomization by the principal investigator only. A separate anesthetist will do a pre-anesthetic checkup.

   Premedication (Oral Midazolam 0.3 mg/kg) will be prescribed. On the day of surgery, the patient will be premedicated; the intravenous cannula will be inserted inward. On arrival of the patients to the operative theatre, ASA monitors will be attached ( ECG, non-invasive blood pressure, and SPO2 ). Anesthesia will be induced with an intravenous agent: Propofol: 2 mg/kg, inhalational anesthesia: sevoflurane, fentanyl 1 mic/kg, glycopyrrolate 10 mics/kg and a supraglottic airway device (Laryngeal mask airway) will be placed. Inhalational agent: Sevoflurane will be continued for the maintenance of anesthesia. The patient will be positioned for the block, and the block will be given as per randomization by one of the two expert pediatric anesthesia consultants following the study protocol. The postoperative nausea and vomit prophylaxis will be given with granisetron : 0.01 mg/kg & Dexamethasone 0.15mg/kg. For multimodal intraoperative analgesia Paracetamol 7.5 mg/kg for < 10 kg weight and 15 mg/kg for > 10 kg weight will be infused intravenously. At the end of the procedure, the anesthesia will be turned off, and the child will be extubated after waking up as per the standard procedure. Then the child will be shifted to PACU (Post-Anesthesia Care Unit).

   For caudal block:

   With the patient in the lateral position, the sacral cornua are identified by palpation using the anatomic landmarks. Sterile skin preparation and draping of the entire region are performed. A high-frequency ultrasound probe is placed in the transverse plane across the two sacral cornua. The sacral cornua can be visualized as two symmetric hyperechoic arches, with a hypoechoic shade underneath both lines, bridging these two structures. An appropriately sized needle is inserted into the space between the two cornua. A distinct "pop" is felt as the needle tip penetrates the sacrococcygeal ligament. At this point, the probe's orientation is changed into the sagittal plane. The caudal canal is identified as a hypoechoic canal tapering off caudally and bordered by dorsal and ventral hyperechoic bands. The dorsal band is formed by the dorsal bony aspect of the caudal canal cranially and the sacrococcygeal ligament caudally. The ventral band is formed by the ventral bony surface of the caudal canal. The needle will be advanced under ultrasound guidance, keeping the tip of the needle in view at all times; the drug will be injected after placement of the needle tip in the caudal space. Levobupivacaine 0.25%, 1 ml/kg will be injected into the space.

   For Ilio-inguinal/iliohypogastric nerve block technique:

   Position the patient supine. Prepare skin with antiseptic. Place the high-frequency ultrasound probe on the anterior abdominal wall along the line joining the anterior superior iliac spine (ASIS) and the umbilicus. The ilioinguinal and iliohypogastric nerves are seen as hypoechoic structures with a hyperechoic border. They lie in the plane between the internal oblique muscle and the transversus abdominis muscle close to the ASIS. Insert the block needle in the plane from medial to lateral and ensure that there is always a good image of the needle tip as the needle is advanced. The dose of levobupivacaine will be 0.4 ml/kg of 0.25% concentration to be deposited slowly around the nerves in the transversus abdominis plane.

   Standard intraoperative ASA monitoring will be done and compared amongst the two groups.

   PACU and Ward:

   During the postoperative time, patients will be transferred to PACU and the ward when they recover from anesthesia and will be observed by trained nurses. FLACC score will be assessed & documented 30 minutes after the end of anesthesia and before discharge from PACU, postoperatively in Ward at 2 Hours, 3 hours, 6 hours from the end of anesthesia, and or at the time of discharge from the ward.

   Follow up at Home:

   The patients will be followed up on days 2 and 7 for pain with a Numeric rating scale (NRS), consumption of analgesics, resumption of daily basic and routine preoperative activities, and any untoward side effects.

   Rescue analgesia:

   Intraoperative rescue analgesia: For inadequate analgesia due to block, rescue analgesia will be provided with morphine 50 mics/kg aliquots.

   Postoperative rescue analgesia:

   PACU: The pain will be assessed by PACU staff and nurses in the ward using the FLACC scale, and rescue analgesia will be given with Morphine 50 mics/kg aliquots (highest 200 mic/kg).

   Ward: In the ward rescue will be with Paracetamol 7.5-10 mg/kg for children< 10 kg and 15 mg/kg for children > 10 kg. The number of times the rescue is given will be recorded.

   Home: Syrup Paracetamol 10 mg/kg sos (when needed) or every 8 hours will be prescribed.

   Complications:
   * Local anesthetic systematic toxicity (LAST)
   * Hemodynamic changes
   * Infection
   * Injury to the nerve roots
   * Subdural injection & Hematoma formation
   * Urinary retention
   * Bleeding

   Troubleshooting:

   Inadequate block or Failed block:

   The depth of the sacral canal at the apex of the sacral hiatus and the length of the sacrococcygeal ligament between the apex of the sacral hiatus and the sacral base is associated with difficulty in performing CEB. In case of failed or inadequate block patient, rescue analgesia will be provided with morphine 50 mics/kg. The pain will be assessed by PACU staff and nurses in the ward using the FLACC scale. In the ward, rescue will be with Paracetamol 15 mg/kg orally.

   Hemodynamic changes:

   Mainly hemodynamic changes are observed immediately after the block, and they are mild. The patients will be continuously monitored during the perioperative period. And any hemodynamic instability will be immediately treated with intravenous fluids and vasopressors if it is significant.

   Bleeding:

   It is rarely encountered. Bleeding can be controlled by putting pressure on the area of direct needle trauma with hematoma formation. The management includes conservative treatment and surgical exploration. Especially if a hematoma forms, it should be removed promptly. Comprehensive knowledge of anatomy and adept skills are crucial to avoid nerve injuries, and that's why experts in this study will perform the blocks.

   LAST:

   It is rare as the blocks are usually ultrasound-guided, and drugs are given in smaller amounts than the toxic levels. They are given with frequent aspirations to prevent injecting into blood vessels. In pediatric practice, early warning signs and symptoms of toxicity may be masked by the concurrent administration of general anesthesia. This means the first sign may be arrhythmia or cardiovascular collapse. Consider the following when managing local anesthetic toxicity:
   * Stop the local anesthetic injection.
   * Institute essential life support and call for assistance.
   * Secure the airway, ventilate with 100% oxygen, and gain intravenous access.
   * Seizures can be managed with a benzodiazepine or anesthetic induction agent.
   * If a cardiac arrest has occurred, commence advanced life support.
   * Note that arrhythmias are often refractory, and resuscitation should therefore be prolonged.
   * Treatment with IntraLipid: An initial dose of 20% lipid emulsion at 1.5 ml/kg or a 100 ml bolus can be administered over a few minutes. This can be repeated after 5 minutes for 2 or more times for persistent hemodynamic instability. The bolus(es) should immediately be followed by a continuous infusion at 0.25-0.5 ml/kg/min.[3] The infusion should run for a minimum of 10 minutes after the return of hemodynamic stability. However, there are documented reports of recurrent systemic toxicity even after this. For this reason, patients should be admitted for at least 12 hours for observation and additional doses of intralipid as needed for rebound symptoms or hemodynamic compromise.12

   Infection:

   It is a rare complication, might be seen after a few days postoperatively, and it will be treated with appropriate antibiotics after postoperative surveillance during the follow-up.

   Injury to nerve roots:

   This is a rare complication, especially so when a block is guided by ultrasound. But in case of a very rare event, it still happens; it usually recovers within a few weeks, and follow-up is required if the recovery is not observed, then the patient will be managed by neurology consultation.

   Subdural injection These complications are rare as the subdural sac is away from caudal space in children. And the blocks in this study will be done with ultrasound guidance. Still, if it occurs, the chance of hemodynamic instability is low as the volume and concentration of local anesthetics will be low (0.25%) for analgesia.

   Urinary retention:

   It is usually transient and improves with regression in the block.

   Roles:

   A statistician will send an age-stratified-computer-generated block randomization sequence to the Principal investigator, who will keep it under lock. The Principal Investigator will allocate the cases according to the computerized randomization sequence received.

   Anesthetist doctor 1 will assess the patient and give anesthesia, perform the block and fill proforma 1 and give the patient a code on proforma 2. There will be 2 anesthetists, well-trained in the block and pediatric anesthesia techniques, will be performing the blocks and giving anesthesia. Anesthetist doctor 2 will do the same procedure next time.

   Assessor 1 will assess the patient in PACU using the FLACC scale 30 minutes after the end of anesthesia and before discharge from PACU. He/She will fill the proforma 2 with the patient code and not the identity.

   Assessor 2 will assess the patient in the ward at 2, 3, and 6 hours and or at discharge from the ward.

   Assessors 1 or 2 will follow up with the patient telephonically at home on days 2 and 7.

   The data entry with patient code on the master chart by the Principal investigator without knowing the patient's identity.

   Data collection:

   The following data will be collected:

   Demographic Data: Age, gender, ASA grading, comorbidities, surgery Lab Data: Routine blood investigations like complete blood count and coagulation profile.

   Anesthesia and block details: Type of airway device, hemodynamic, block details: block name, normal/abnormal anatomy, local anesthetics injected; rescue analgesics needed, FLACC score at 30 minutes after arrival and before discharge from PACU, postoperatively in Ward at 2 Hours, 3 hours, 6 hours and or at time of discharge from the ward and at home on day 2 and day 7.

   The recorded patient data with code and no name will be entered by one of the assigned co-investigators into the password-protected master chart.

   Pain assessment: FLACC score will be assessed & documented 30 minutes after arrival and before discharge from PACU, postoperatively in Ward at 2 Hours, 3 hours, 6 hours, and or at the time of discharge. Our target FLACC score is 1-3. Whereas pain assessment at home will be done with a numeric rating scale (NRS).

   Justification of the current study:

   This study will help to identify a more effective analgesia technique for common pediatric inguinal surgeries. These nerve block techniques are safe and have been in use already but not evaluated. Hence, this will be a valuable study to evaluate analgesia efficacy as well as a reduction in the use of rescue analgesics, thereby avoiding the side effects of rescue analgesics. Not only effectiveness, but we will also study the time of discharge and resumption of independent activities. The better-found technique may help enhance recovery after surgery (ERAS) for this patient population.

   ETHICAL REVIEW:

   After getting ethical approval and a Clinicaltrials registry, an appropriate population of patients will be approached. A proper explanation will be done with the help of a patient information sheet in the local and English languages. Informed consent will be obtained before randomization from parents. Patient confidentiality will be maintained strictly. All Proforma and Consent forms will be kept under lock and key. The master chart will not carry patient names, and even MRN will not be accessible to anyone except the principal investigator. In the end, the study subjects will be given code numbers in the final master chart, and their ID will not be revealed to the statistician. An interim analysis will be done to assess the results then continuation with the study will be decided after 25% of the cases on each arm.

   Data Management and Analyses:

   Statistical Method The null hypothesis for the primary endpoint is that the analgesic effect between the two blocks is not different. The alternative hypothesis is that the block has different analgesic efficacy, measured in terms of pain score (FLACC and NRS). The hypothesis will be two-sided and tested at the 5% significance level.

   Demographics and baseline characteristics will be summarized. Summary of continuous variables will be presented using N, Mean, Standard Error of mean (SE), Standard Deviation (SD), Median and Range (Minimum and Maximum), and interquartile ranges (IQR). The categorical variables will be presented using numbers and percentages. A Student's t-test will be applied for primary and secondary endpoints of continuous variables to test the mean difference between the groups. The t-test will be tested as two-sided hypotheses at a 5% significance level. Treatment differences will be confirmed and considered significant if the p-value reported is < 0.05. The presentation of results from a statistical analysis using a t-test will include the estimated mean difference between the groups for endpoint values. Continuous variables with non-normal distribution will also be analyzed using the Mann-Whitney test. The Hodges-Lehmann estimate and 95% confidence interval for the median difference will be presented along with p-values using the Mann-Whitney test. Dichotomous or nominal categorical variables were analyzed by either the Pearson Chi-square or Fisher's exact test. Disposition of patients (subject screened, randomized, and disposition at the end of study along with reasons for withdrawals) in the study will be summarized as the number of subjects and percentage.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 12 years
* ASA I and II
* Type of surgery (Inguinal surgeries)

Exclusion Criteria:

* Refusal of consent
* ASA III and higher risk group
* Hemodynamically unstable
* Local infection over the insertion site
* Coagulopathy
* Known allergy to Local Anaesthetic medications
* Difficult anatomy

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Degree of pain relief | upto 1-2 days
  Degree of analgesia will be checked postoperatively at 30 minutes after anesthesia in PACU, postoperatively in ward at 2, 3 and 6 hours from end of anesthesia and or at time of discharge from ward whichever is earlier.

SECONDARY OUTCOMES:
Change in use of rescue analgesia postoperatively | upto 1-2 days
  Change in use of rescue analgesia postoperatively till period of discharge from the ward

OTHER OUTCOMES:
Postoperative length of stay | upto 1-2 days
  Postoperative length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Burad, MD, EDIC, Principal Investigator — Sultan Qaboos University Hospital
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after completion and publication of the study on Mendeley
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the Publication of the study, the data will be available on Mendeley for a few years
Access Criteria: Any researcher requesting the data for further research will be given access.
URL: http://data.mendeley.com/

REFERENCES:
- [Background] Finley AG, McGrath PJ, Forward PS, McNeill G, Fitzgerald P. Parents' management of children's pain following 'minor' surgery. Pain. 1996 Jan;64(1):83-87. doi: 10.1016/0304-3959(95)00091-7. PMID 8867249
- [Background] Rawal N, Sjostrand U, Christoffersson E, Dahlstrom B, Arvill A, Rydman H. Comparison of intramuscular and epidural morphine for postoperative analgesia in the grossly obese: influence on postoperative ambulation and pulmonary function. Anesth Analg. 1984 Jun;63(6):583-92. PMID 6233917
- [Background] Dalens B, Hasnaoui A. Caudal anesthesia in pediatric surgery: success rate and adverse effects in 750 consecutive patients. Anesth Analg. 1989 Feb;68(2):83-9. PMID 2913854
- [Background] Disma N, Tuo P, Pellegrino S, Astuto M. Three concentrations of levobupivacaine for ilioinguinal/iliohypogastric nerve block in ambulatory pediatric surgery. J Clin Anesth. 2009 Sep;21(6):389-93. doi: 10.1016/j.jclinane.2008.10.012. PMID 19833270
- [Background] Dawes JM, Cooke EM, Hannam JA, Brand KA, Winton P, Jimenez-Mendez R, Aleksa K, Lauder GR, Carleton BC, Koren G, Rieder MJ, Anderson BJ, Montgomery CJ. Oral morphine dosing predictions based on single dose in healthy children undergoing surgery. Paediatr Anaesth. 2017 Jan;27(1):28-36. doi: 10.1111/pan.13020. Epub 2016 Oct 25. PMID 27779356
- [Background] Dua A, Afzal M. Caudal Anesthesia. 2025 Feb 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK551693/ PMID 31869157
- See also: Nysora website — https://www.nysora.com/techniques/neuraxial-and-perineuraxial-techniques/caudal-anesthesia/
- See also: ilioinguinal block complications — http://www.openanesthesia.org/aba_ilioinguinal_block_-_complications/
- See also: Nysora: local anesthetic systemic toxicity — http://www.nysora.com/topics/complications/local-anesthetic-systemic-toxicity/
- See also: ilioinguinaliliohypogastric-block — https://www.euroespa.com/science-education/specialized-sections/espa-pain-committee/us-regional-anaesthesia/truncal-blocks/ilioinguinaliliohypogastric-block
- See also: Dosing-guidelines-for-pediatric-procedural-sedation-and-analgesia — https://www.medscape.com/answers/109695-177728/what-are-the-dosing-guidelines-for-pediatric-procedural-sedation-and-analgesia-psa
- See also: Role-of-fentanyl-in-pediatric-sedation — https://www.medscape.com/answers/804045-188308/what-is-the-role-of-fentanyl-in-pediatric-sedation